CLINICAL TRIAL: NCT00211081
Title: Impact of Spironolactone on Endothelial Function in Patients With Single Ventricle Heart
Brief Title: Spironolactone in Patients With Single Ventricle Heart
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, William T. Mahle, MD, Principal Investigator, Emory University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0954-2004
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Results first posted 2014-12-16 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-10

CONDITIONS: Congenital Disorders
Keywords: Congenital Heart Disease; Spironolactone; >17 years old; undergone Fontan procedure; endothelial function
MeSH Terms: conditions — Congenital, Hereditary, and Neonatal Diseases and Abnormalities; Heart Defects, Congenital | interventions — Spironolactone; Pharmaceutical Preparations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Open Label (Experimental)
  Interventions: Drug: Spironolactone (drug)

INTERVENTIONS:
Drug: Spironolactone (drug) — 1 mg/kg/day; afer 2 weeks doubled to 2/mg/kg/day. Patient's with endothelium-dependent brachial artery vasodilation and single-ventricle should show improvement within 4-8 weeks. Patients and their labs who are receiving Spironolactone will be followed.

SUMMARY:
Ultrasound is a technique that can provide images of the blood vessels such as arteries. The size of the arteries, such as the main blood vessel in the arm, can change under different conditions. Using ultrasound we can see how arteries change with movement or even drugs. We want to use ultrasound to see how blood vessels look in patients with Congestive Heart Failure (CHF) and to also see how a drug called Spironolactone, commonly prescribed for patients with this disease, effects blood vessel function in patients with congestive heart failure. This information may be used to change the standard of care for patients with heart failure especially if we show that Spironolactone has a positive effect on vessel function in patients with CHF.

DETAILED DESCRIPTION:
Spironolactone The starting dose of spironolactone is 1 mg/kg/day. After two weeks this dose will be doubled to the same maximum dose (2/mg/kg/day) as in RALES. If side effects occur or plasma urea and electrolytes became deranged the dose will be halved. Patients unable to tolerate the minimum dose will be withdrawn. Measurement of serum electrolytes will occur at baseline, at two weeks, and at time of repeat evaluation.

Endothelial Function

Subjects with single ventricle will have an evaluation of endothelial function:

1. At baseline
2. On spironolactone- 4-5 weeks after initial study.

Imaging protocol:

The diameter of the brachial artery will be measured from two-dimensional ultrasound images, using a 12 MHz linear array transducer and an Accuson Sequoia system (Accuson, Mountainview, California). Measurements of the brachial artery will be obtained:

1. In a resting state
2. During limb ischemia
3. In response to reactive hyperemia
4. At rest

Reactive hyperemia will be induced by inflating a standard blood pressure cuff to 50 mm Hg above the systolic blood pressure for 4.5 minutes and then deflating the cuff.

After data collection, the DICOM-formatted images will be transferred to a PC for investigator-blinded measurement of brachial artery diameter using image analysis software (Brachial Tools 3.1, Medical Imaging Applications, Iowa).

Measurement of prognostic markers:

Blood samples

Plasma beta-type natriuretic peptide, form assay, TNF alpha and a Cytokine panel will be drawn at base line and at the final 4-5 week visit for this study.

Samples will be collected between 11 am and 1 pm after 30 minutes' supine rest. The samples will be centrifuged and plasma stored at -70°C (peptides) or -20°C (other samples). Plasma [beta]-type natriuretic peptide (BNP) samples will be collected into EDTA and aprotonin and measured by radioimmunoassay 6-minute walk test.

A 6-minute walk test will be performed at the first visit and the last visit. During this test, signs and symptoms will be recorded (i.e. chest pain and shortness of breath) to determine toleration of daily activity. A doctor or nurse will conduct this test and the patient will be provided the opportunity to stop or rest if symptoms become severe.

Outcome measures

The primary outcome measure will be the change in flow mediated dilation (during reactive hyperemia). This will be expressed as a percentage.

Secondary outcome measures will include changes in BNP, Form assay, TNF alpha, Cytokine panels and the 6-minute walk test.

Statistical analysis

We and others have previously shown that asymptomatic patients with the Fontan operation have a mean flow-mediated dilation of approximately 4% compared to 8-9% in controls. In order to detect a 25% change in FMD, with a power of 0.80, the current study would require a patient population of 13 cases. There are currently over 40 patients with single ventricle who are followed in the adult congenital clinic at Emory University.

We plan on enrolling 20 patients into this study.

ELIGIBILITY:
Inclusion Criteria:

* Single Ventricle Subjects
* >17 years
* have undergone Fontan Procedure

Exclusion Criteria:

* History of smoking
* Diabetes mellitus
* Renal failure (serum creatinine > 2.5 mg/dl)
* Recovering spironolactone for maintenance therapy
* History of hyperkalemia (serum potassium> 5.5 mEq/L)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2004-11; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William T Mahle, MD, Principal Investigator — Emory University; Arshed Quyyumi, MD, Principal Investigator — Emory University; Wendy M Book, MD, Principal Investigator — Emory University; Michael E McConnell, MD, Principal Investigator — Emory University
Locations (1):
- Emory Clinic, Atlanta, Georgia, United States

REFERENCES:
- [Background] Celermajer DS, Sorensen KE, Gooch VM, Spiegelhalter DJ, Miller OI, Sullivan ID, Lloyd JK, Deanfield JE. Non-invasive detection of endothelial dysfunction in children and adults at risk of atherosclerosis. Lancet. 1992 Nov 7;340(8828):1111-5. doi: 10.1016/0140-6736(92)93147-f. PMID 1359209
- [Background] Sorensen KE, Celermajer DS, Spiegelhalter DJ, Georgakopoulos D, Robinson J, Thomas O, Deanfield JE. Non-invasive measurement of human endothelium dependent arterial responses: accuracy and reproducibility. Br Heart J. 1995 Sep;74(3):247-53. doi: 10.1136/hrt.74.3.247. PMID 7547018
- [Background] Celermajer DS. Endothelial dysfunction: does it matter? Is it reversible? J Am Coll Cardiol. 1997 Aug;30(2):325-33. doi: 10.1016/s0735-1097(97)00189-7. PMID 9247501
- [Background] Celermajer DS, Sorensen K, Ryalls M, Robinson J, Thomas O, Leonard JV, Deanfield JE. Impaired endothelial function occurs in the systemic arteries of children with homozygous homocystinuria but not in their heterozygous parents. J Am Coll Cardiol. 1993 Sep;22(3):854-8. doi: 10.1016/0735-1097(93)90203-d. PMID 8354824
- [Background] Anderson TJ, Elstein E, Haber H, Charbonneau F. Comparative study of ACE-inhibition, angiotensin II antagonism, and calcium channel blockade on flow-mediated vasodilation in patients with coronary disease (BANFF study). J Am Coll Cardiol. 2000 Jan;35(1):60-6. doi: 10.1016/s0735-1097(99)00537-9. PMID 10636260
- [Background] Gidding SS, Rocchini AP, Moorehead C, Schork MA, Rosenthal A. Increased forearm vascular reactivity in patients with hypertension after repair of coarctation. Circulation. 1985 Mar;71(3):495-9. doi: 10.1161/01.cir.71.3.495. PMID 3971523
- [Background] Yang SG, Rychik J. Mesenteric blood flow patterns: A link to protein-losing enteropathy after the Fontan operation. Circulation 1999;100-18:A3583.

RESULTS

PARTICIPANT FLOW:
Groups:
- Spironolactone: Subjects took spironolactone at 25 mg daily. After two weeks, Spironolactone was doubled to 50 mg daily for remaining 2 weeks.
Period: Overall Study
Arm/Group | Spironolactone
Started | 12
Completed | 10
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Spironolactone
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3
  Between 18 and 65 years | 9
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 28 [15 to 42]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 7
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Change in Flow Mediated Dilation
Description: Flow-mediated dilation of the brachial artery will be measured using high-resolution ultrasound. Arterial diameter will be measured above the small cavity in the elbow joint from ultrasound images at rest in response to an increase in blood flow to the area.
Time Frame: Baseline, Post-Intervention (4 Weeks)
Population: Subjects that completed all study visits.
Measure: Mean (Standard Deviation); unit: Percentage of brachial artery diameter
Arm/Group | Spironolactone
Number analyzed (Participants) | 10
Percentage of brachial artery diameter | 5.5 (2.1)

2. Secondary Outcome: C-Reactive Protein Level
Description: The normal reference range for C-reactive protein is as follows: CRP: 0-10mg/L
Time Frame: Baseline, Post-Intervention (4 Weeks)
Population: Subjects that completed all study visits.
Measure: Median (Inter-Quartile Range); unit: mg/L
Arm/Group | Spironolactone
Number analyzed (Participants) | 10
mg/L
  Baseline | 1.10 [.15 to 21.4]
  4 Week Follow Up | 1.10 [.17 to 19.95]

3. Secondary Outcome: Interleukin-6 (IL-6) Level
Description: The normal result for IL-6 for Interleukin 6 is < 5pg/ml.
Time Frame: Baseline, Post-Intervention (4 Weeks)
Population: Subjects that completed all study visits.
Measure: Median (Inter-Quartile Range); unit: pg/ml
Arm/Group | Spironolactone
Number analyzed (Participants) | 10
pg/ml
  Baseline | 1.96 [1.18 to 14.78]
  4 Week Follow Up | 1.54 [1.29 to 5.29]

4. Secondary Outcome: Interleukin 1 Beta (IL1b) Level
Description: The normal result for IL1b is <3.9 pg/mL.
Time Frame: Baseline, Post-Intervention (4 Weeks)
Population: Subjects that completed all study visits.
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Spironolactone
Number analyzed (Participants) | 10
pg/mL
  Baseline | .38 [.23 to .53]
  4 Week Follow Up | .23 [.08 to .48]

5. Secondary Outcome: Interleukin-10 (IL10) Level
Description: The normal result for IL-10 for Interleukin 10 is < 18pg/ml.
Time Frame: Baseline, Post-Intervention (4 Weeks)
Population: Subjects that completed all study visits.
Measure: Median (Inter-Quartile Range); unit: 18pg/ml
Arm/Group | Spironolactone
Number analyzed (Participants) | 10
18pg/ml
  Baseline | .26 [.10 to .36]
  4 Week Follow Up | .13 [.10 to .70]

6. Secondary Outcome: Tumor Necrosis Factor-Alpha (TNF-a) Level
Description: The normal result for TNF-a is <5.6 pg/mL.
Time Frame: Baseline, Post-Intervention (4 Weeks)
Population: Subjects that completed all study visits.
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Spironolactone
Number analyzed (Participants) | 10
pg/mL
  Baseline | 2.20 [1.17 to 5.72]
  4 Week Follow Up | 2.42 [1.54 to 5.94]

7. Secondary Outcome: Change in 6 Minute Walk Test Score
Time Frame: Baseline, Post-Intervention (4 Weeks)
Population: This assessment was not completed during the study.
Arm/Group | Spironolactone
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected throughout the duration of the study (4 years).
Arm/Group | Spironolactone
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No